CLINICAL TRIAL: NCT04600284
Title: A Randomized, Open Label, Multiple Dose, Crossover Study to Evaluate Drug-drug Interaction of AD-2101 and AD-2102 in Healthy Male Subjects
Brief Title: Evaluating the Pharmacokinetic Interaction Between AD-2101 and AD-2102
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Addpharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AD-210DDI
Record Dates: First submitted 2020-10-19; First posted 2020-10-23 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Sequence 1 (Experimental): Period 1: AD-2101 Period 2: AD-2102 Period 3: AD-2101 + AD-2102
  Interventions: Drug: AD-2101; Drug: AD-2102; Drug: AD-2101 + AD-2102
- Sequence 2 (Experimental): Period 1: AD-2101 Period 2: AD-2101 + AD-2102 Period 3: AD-2102
  Interventions: Drug: AD-2101; Drug: AD-2102; Drug: AD-2101 + AD-2102
- Sequence 3 (Experimental): Period 1: AD-2102 Period 2: AD-2101 Period 3: AD-2101 + AD-2102
  Interventions: Drug: AD-2101; Drug: AD-2102; Drug: AD-2101 + AD-2102
- Sequence 4 (Experimental): Period 1: AD-2102 Period 2: AD-2101 + AD-2102 Period 3: AD-2101
  Interventions: Drug: AD-2101; Drug: AD-2102; Drug: AD-2101 + AD-2102
- Sequence 5 (Experimental): Period 1: AD-2101 + AD-2102 Period 2: AD-2101 Period 3: AD-2102
  Interventions: Drug: AD-2101; Drug: AD-2102; Drug: AD-2101 + AD-2102
- Sequence 6 (Experimental): Period 1: AD-2101 + AD-2102 Period 2: AD-2102 Period 3: AD-2101
  Interventions: Drug: AD-2101; Drug: AD-2102; Drug: AD-2101 + AD-2102

INTERVENTIONS:
Drug: AD-2101 — AD-2101 16/5mg
Drug: AD-2102 — AD-2102 25mg
Drug: AD-2101 + AD-2102 — AD-2101 16/5mg + AD-2102 25mg

SUMMARY:
The purpose of this study is to evaluate the Pharmacokinetic Interaction Between AD-2101 and AD-2102 in healthy male subjects.

DETAILED DESCRIPTION:
To evaluate the pharmacokinetic Interaction, safety and tolerability of the combination compared with the administration of AD-2101 and AD-2102.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male between 19 and 50 years of age at the time of screening
* Weight above 50 kg and body mass index (BMI) between 17.5 kg/m2 and 30.5 kg/m2

Exclusion Criteria:

* Clinically significant disease or history of clinically significant disease such as cardiovascular, respiratory, liver, kidney, digestive, hematologic/oncologic, endocrine, immunologic, urinary, psychiatric
* Gastrointestinal problem or history of gastrointestinal problem and history of gastrointestinal surgery
* A person who has a history of drug abuse
* AST, ALT, Total bilirubin values over than 2 times of UNL at screening
* Creatinine clearance under 80mL/min

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration | pre-dose to 24 hours
  Cmax,ss of the total ingredient of AD-2101 and AD-2102
Area under the plasma concentration versus time curve | pre-dose to 24 hours
  AUCt,ss of the total ingredient of AD-2101 and AD-2102

SECONDARY OUTCOMES:
Time to reach Cmax | pre-dose to 24 hours
  Tmax,ss of the total ingredient of AD-2101 and AD-2102
Clearance | pre-dose to 24 hours
  CLss/F of the total ingredient of AD-2101 and AD-2102
Bottom Plasma Concentration | pre-dose to 24 hours
  Cmin,ss of the total ingredient of AD-2101 and AD-2102
Number of participants with adverse events | From Day 1 up to Day 66
  Incidence rate of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: HyeWon Chung, Principal Investigator — Korea University Guro Hospital
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea